CLINICAL TRIAL: NCT07334782
Title: Investigation of the Effects of Vertebral Axial Loading Walking Training Added to Core Stabilization Exercises on Pain, Trunk Sensory Function, Muscle Strength and Endurance, Balance, and Proprioception in Patients With Chronic Low Back Pain
Brief Title: Effects of Vertebral Axial Loading Walking Combined With Core Stabilization Exercises in Individuals With Chronic Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nilay Kalender, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTREK24/69
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Chronic Low Back Pain; Core Stabilization Exercise; Spinal Stabilization; Proprioception; Sensorimotor Control; Physiotherapy Rehabilitation; Neuromuscular Control; Vertebral Axial Loading; Balance; Trunk Muscle Strength; Trunk Muscle Endurance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stabilization Exercises plus Vertebral Axial Loading Walking Training (CSE+ALWT Group) (Experimental): Participants in this group receive a standardized core stabilization exercise program combined with vertebral axial loading proprioceptive walking training. The intervention is supervised by a physiotherapist and applied three sessions per week for six weeks.
  Interventions: Behavioral: Core Stabilization Exercises Plus Vertebral Axial Loading Walking Training
- Core Stabilization Exercises Only (CSE Group) (Active Comparator): Participants in this group receive the standardized core stabilization exercise program alone, supervised by a physiotherapist, three sessions per week for six weeks.
  Interventions: Behavioral: Exercise - Core Stabilization Exercise Program

INTERVENTIONS:
Behavioral: Exercise - Core Stabilization Exercise Program — Participants receive a physiotherapist-supervised core stabilization exercise program applied three sessions per week for six weeks. Before training, participants are educated about core muscle function and taught the abdominal bracing maneuver. Exercises are performed with neutral spinal alignment and controlled diaphragmatic breathing. Each session includes warm-up and cool-down exercises. The program consists of deep abdominal muscle activation, lower extremity movements with maintained trunk stability, bridging exercises, modified curl-up, and quadruped stabilization exercises. Exercises are demonstrated by the physiotherapist, performed with progressive repetitions, and corrected using verbal and manual feedback. The training is supervised by a physiotherapist and applied three sessions per week for six weeks.
  Arms: Core Stabilization Exercises Only (CSE Group)
Behavioral: Core Stabilization Exercises Plus Vertebral Axial Loading Walking Training — Participants receive the same core stabilization exercise program combined with vertebral axial loading proprioceptive walking training. Axial loading is applied through the vertex of the head using external weights ranging from 50 to 250 grams, adjusted according to individual tolerance. Walking is performed at a constant slow pace using a metronome set at 72 beats per minute. The initial walking distance is 40 meters and is progressively increased by 20 meters per week, reaching up to 140 meters. The intervention is supervised by a physiotherapist and applied three sessions per week for six weeks.
  Arms: Core Stabilization Exercises plus Vertebral Axial Loading Walking Training (CSE+ALWT Group)

SUMMARY:
Chronic low back pain is a common musculoskeletal condition persisting for more than three months and is associated with pain, functional limitations, impaired balance, altered proprioception, reduced trunk muscle performance, and decreased quality of life. Previous studies have demonstrated that individuals with chronic low back pain exhibit altered sensory input from spinal structures and impaired neuromuscular control, which may contribute to persistent pain and movement dysfunction. Although exercise-based physiotherapy approaches, particularly core stabilization exercises, are widely recommended and effective in the management of chronic low back pain, sensory deficits related to balance, proprioception, and body awareness are often insufficiently addressed in conventional rehabilitation programs.

Vertebral axial loading walking training is a functional rehabilitation approach involving slow, controlled walking under gentle vertical loading applied along the spinal axis. This intervention is thought to enhance afferent sensory input from spinal mechanoreceptors, potentially improving balance control, proprioception, and motor coordination. This randomized controlled study aims to investigate the effects of adding vertebral axial loading walking training to a standard core stabilization exercise program on pain intensity, balance, proprioception, trunk muscle strength and endurance, and body awareness in individuals with chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain is one of the leading causes of disability worldwide and is characterized not only by persistent pain but also by impairments in postural control, proprioception, trunk muscle function, and body awareness. Neurophysiological studies have demonstrated that individuals with chronic low back pain exhibit altered afferent input from lumbar spinal structures and changes in central nervous system processing, resulting in impaired sensorimotor control and delayed trunk muscle activation. These alterations may negatively affect balance, movement coordination, and functional performance, thereby contributing to the chronicity of symptoms. Core stabilization exercises are commonly prescribed to improve trunk muscle strength, endurance, and neuromuscular control and have demonstrated beneficial effects in individuals with chronic low back pain. However, evidence suggests that traditional exercise programs may not sufficiently stimulate sensory receptors involved in proprioceptive input and postural regulation. Impaired proprioception and reduced body awareness have been identified as key factors associated with ongoing pain and functional limitations in this population. Vertebral axial loading walking training is a novel and functional intervention that applies gentle vertical loading along the spinal axis during slow and controlled walking. Axial loading is thought to stimulate spinal mechanoreceptors and enhance sensory feedback, thereby facilitating improved proprioceptive awareness, postural stability, and motor coordination during functional activities. This approach is practical, cost-effective, and easily integrated into rehabilitation settings. In this randomized controlled study, participants with chronic low back pain will be allocated to either a core stabilization exercise program alone or a combined intervention consisting of core stabilization exercises and vertebral axial loading walking training. Outcome measures will include pain intensity, balance performance, lumbar proprioception, trunk muscle strength and endurance, and body awareness. Assessments will be conducted at baseline and after the intervention period. The results of this study are expected to provide evidence for a more comprehensive rehabilitation strategy by integrating sensory-based and functional axial loading approaches into physiotherapy programs for individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 55 years
* Able to read and write
* Not using regular medication during the study period
* Voluntary participation and willingness to comply with study procedures

Exclusion Criteria:

* Presence of lumbar radiculopathy or neurological deficits
* Presence of specific spinal pathologies, including scoliosis, kyphosis, malignancy, fracture, infection, or inflammatory joint or bone diseases
* Presence of major or chronic systemic diseases, including diabetes mellitus, rheumatoid arthritis, or systemic lupus erythematosus
* Presence of any neurological disease, such as stroke, Parkinson's disease, or multiple sclerosis
* Presence of any condition affecting balance, including cerebellar ataxia, vertigo, Ménière's disease, inner ear labyrinthitis, or vestibular neuritis
* History of spinal surgery
* History of minimally invasive spinal procedures or injections, including platelet-rich plasma (PRP), growth factor-rich plasma (GFRP), corticosteroids, or other pharmacological injections
* History of major lower extremity surgery, including knee arthroplasty, hip arthroplasty, high tibial osteotomy, or meniscal surgery
* Presence of lower extremity musculoskeletal injuries, including meniscal or ligament injuries or chronic ankle instability
* Presence of lower extremity deformities, including talipes equinovarus, genu varum, genu valgum, or coxa vara/valga
* Presence of cognitive impairment or diagnosed psychiatric disorders
* Pregnancy or being less than 6 months postpartum
* History of cancer or ongoing cancer treatment
* Illiteracy
* Failure to attend three consecutive treatment sessions
* Receipt of physical therapy or rehabilitation within the past 6 months

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Lumbar Proprioception (Active Joint Position Sense) After 6 Weeks of Intervention | Baseline and 6 weeks
  Lumbar proprioception will be assessed by measuring active joint position sense during trunk flexion, lateral flexion, and extension using MATLAB-based angle analysis. The absolute angular error (in degrees) between the target position and the reproduced position will be calculated. Angular error is recorded in degrees, starting from 0° upward. Lower values indicate better proprioceptive accuracy. Higher values indicate impaired proprioception.
Change from Baseline in Pain Intensity at Rest and During Activity After 6 Weeks | Baseline and 6 weeks
  Pain intensity will be assessed using the Numeric Rating Scale (NRS). The scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Lower scores indicate less pain.
Change from Baseline in Lumbar Pressure Pain Threshold After 6 Weeks | Baseline and 6 weeks
  Pressure pain threshold will be measured using a handheld algometer (Algometer commander, JTech Medical) and recorded in kg/cm². Higher values indicate greater pain tolerance, while lower values indicate increased pain sensitivity.
Change from Baseline in Trunk and Hip Muscle Strength After 6 Weeks | Baseline and 6 weeks
  Isometric muscle strength of trunk and hip muscles will be assessed using a digital hand-held dynamometer (Lafeyette Instrument®, Lafayette, IN) during maximal voluntary isometric contraction. Strength values are recorded in Newtons (N) or kilograms (kg). Higher values indicate greater muscle strength

SECONDARY OUTCOMES:
Change from Baseline in Balance Performance Assessed by the Fullerton Advanced Balance Test After 6 Weeks | Baseline and 6 weeks
  Balance performance will be assessed using the Fullerton Advanced Balance Test (FAB-T), consisting of 10 functional balance tasks. Total scores range from 0 to 40. Higher scores indicate better balance performance. Scores ≤25 indicate increased risk of falls.
Change from Baseline in Functional Disability Assessed by the Oswestry Disability Index After 6 Weeks | Baseline and 6 weeks
  Functional disability related to low back pain will be assessed using the Oswestry Disability Index (ODI), version 2.1a.
  Scores range from 0% to 100%, where:
  0% = no disability 100% = maximum disability Higher scores indicate greater disability.
Change from Baseline in Postural Alignment Assessed by the New York Posture Rating Scale After 6 Weeks | Baseline and 6 weeks
  Postural alignment will be evaluated using the New York Posture Rating Scale (NYPRS) based on observational assessment of body segments. Scores range from 0 to 100. Higher scores indicate better postural alignment.
Change from Baseline in Kinesiophobia Assessed by the Tampa Scale of Kinesiophobia After 6 Weeks | Baseline and 6 weeks
  Fear of movement will be assessed using the Tampa Scale of Kinesiophobia (TSK). Total scores range from 17 to 68, with higher scores indicating greater fear of movement. Scores above 37 indicate high levels of kinesiophobia.
Change from Baseline in Health-Related Quality of Life Assessed by the EQ-5D-5L After 6 Weeks | Baseline and 6 weeks
  Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) and the EQ Visual Analogue Scale (EQ-VAS). The EQ-VAS ranges from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. Higher scores indicate better perceived health-related quality of life.
Change from Baseline in Lumbar Range of Motion After 6 Weeks | Baseline and 6 weeks
  Lumbar range of motion was assessed using a 360-degree universal goniometer, which is designed to measure joint position and range of motion across nearly all body joints. The goniometer used in this study was a plastic, full-circle (360°) universal goniometer, allowing continuous angular measurement throughout the full range of motion. Lumbar movements including trunk flexion, extension, right lateral flexion, and left lateral flexion were measured in degrees following standardized assessment procedures. Higher angle values indicate greater lumbar mobility, whereas lower values indicate reduced range of motion.
Change from Baseline in Trunk Muscle Endurance After 6 Weeks | Baseline and 6 weeks
  Trunk muscle endurance will be assessed using the Biering-Sorensen Test for trunk extensor muscles and the Kraus-Weber Test for trunk flexor muscles. Participants will be instructed to maintain the standardized test position for as long as possible, and endurance time will be recorded in seconds, with a maximum duration of 240 seconds. Longer holding times indicate greater trunk muscle endurance.
Change from Baseline in Trunk Sensory Function After 6 Weeks | Baseline and 6 weeks
  Trunk sensory function will be assessed at the L1, L3, and L5 levels using a standardized sensory test battery including light touch sensation, vibration sense, two-point discrimination, and graphesthesia. Light touch sensation will be evaluated using Semmes-Weinstein monofilaments, vibration sense using a 128-Hz tuning fork, two-point discrimination using an aesthesiometer, and graphesthesia by letter recognition tasks applied to the skin. Sensory outcomes will be quantified as tactile threshold (g/mm²), vibration perception time (seconds), minimal two-point discrimination distance (millimeters), and graphesthesia accuracy score, respectively. Lower tactile thresholds, longer vibration perception times, smaller discrimination distances, and higher graphesthesia accuracy indicate better sensory function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations and because the study is conducted as part of a graduate thesis. Aggregated data may be reported in publications.

REFERENCES:
- [Background] Suh JH, Kim H, Jung GP, Ko JY, Ryu JS. The effect of lumbar stabilization and walking exercises on chronic low back pain: A randomized controlled trial. Medicine (Baltimore). 2019 Jun;98(26):e16173. doi: 10.1097/MD.0000000000016173. PMID 31261549
- [Background] Hlaing SS, Puntumetakul R, Khine EE, Boucaut R. Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 30;22(1):998. doi: 10.1186/s12891-021-04858-6. PMID 34847915
- [Background] Bento TPF, Genebra CVDS, Maciel NM, Cornelio GP, Simeao SFAP, Vitta A. Low back pain and some associated factors: is there any difference between genders? Braz J Phys Ther. 2020 Jan-Feb;24(1):79-87. doi: 10.1016/j.bjpt.2019.01.012. Epub 2019 Feb 13. PMID 30782429
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421